CLINICAL TRIAL: NCT03733951
Title: An Open-Label, Multicenter, Dose-Escalation and Expansion Phase Ia/Ib Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of KN046 Monotherapy in Subjects With Advanced Solid Tumors and Lymphoma
Brief Title: KN046 in Subjects With Advanced Solid Tumors and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KN046-CHN-001
Record Dates: First submitted 2018-10-31; First posted 2018-11-07 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumors; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KN046 (Experimental)
  Interventions: Drug: KN046

INTERVENTIONS:
Drug: KN046 — Phase Ia：Intravenous (IV) infusions, 1,3 and 5 milligrams per kilogram (mg/kg) every 2 weeks.
  Phase Ib：Intravenous (IV) infusions, 1 ,3 or 3, 5 milligrams per kilogram (mg/kg) every 2 weeks, the dose of phase Ib based on the result of phase Ia.

SUMMARY:
This is a phase Ia/Ib, open-label, multicenter, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and anti-tumor activity of KN046 in subjects with advanced solid tumors and lymphoma .

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent; willing and able to complete all required procedures of study.
2. With advanced-stage or metastatic tumor (unresectable) and experienced progression since last anti-tumor treatment; standard therapy is not available or rejected.
3. Subjects must have at least one measurable lesion in advanced solid tumors, at least one measurable or assessable lesion in NK/T cell lymphoma.
4. ECOG performance status of 0 or 1.
5. Subject must have adequate organ function.
6. Female patients and males with partners of childbearing potential should be using highly effective contraceptive measures (failure rate of less than 1% per year). Contraception should be continued for a period of 24 weeks after dosing has been completed.
7. Ability to comply with treatment, procedures and PK sample collection and the required study follow-up procedures.

Exclusion Criteria:

1. Known brain metastasis or other CNS metastasis that is either symptomatic or untreated.
2. Is currently participating or has participated in a study of an investigational drug within 4 weeks prior to the first dose of trial treatment.
3. Patients who have received immune checkpoint proteins/antibody/medicine (including PD-1, PD-L1, etc) for treatment.
4. Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management.
5. Subjects with active autoimmune diseases or history of autoimmune diseases should be excluded.
6. Active HBV or HCV infection.
7. Known HIV infection or known history of acquired immune deficient syndrome (AIDS).
8. Any unresolved CTCAE Grade ≥ 2 toxicities from prior anti-cancer therapy with the exception of vitiligo, alopecia.
9. Patients who have serious hypersensitive reaction to monoclonal antibodies, and have history of uncontrolled allergic asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
In the dose escalation part, number of participants with dose limiting toxicity (DLT). | During the first 4 weeks of treatment.
In the dose expansion part,Objective response rate (ORR). | up to 2 years.
  Objective response is defined as complete response (CR) or partial response (PR)
In the dose expansion part, Duration of response (DoR). | up to 2 years.
  Duration of response is defined as the time period from the date of initial independent review committee assessed CR or PR until the date of PD or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - LINYI Cancer Hospital, Linyi, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Chengdu Seventh People's Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Ma Y, Xue J, Zhao Y, Zhang Y, Huang Y, Yang Y, Fang W, Guo Y, Li Q, Ge X, Sun J, Zhang B, Zhang Y, Xiao J, Zhang L, Zhao H. Phase I trial of KN046, a novel bispecific antibody targeting PD-L1 and CTLA-4 in patients with advanced solid tumors. J Immunother Cancer. 2023 Jun;11(6):e006654. doi: 10.1136/jitc-2022-006654. PMID 37263673